CLINICAL TRIAL: NCT01916005
Title: Diagnostic Value of 18F-fluorodeoxyglucose Positron Emission Tomography/Computed Tomography in Prosthetic Valve Endocarditis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2013-A00056-39; 2013-01 (Other: AP HM)
Record Dates: First submitted 2013-05-22; First posted 2013-08-05 (Estimated); Last update posted 2023-04-24 (Actual); Status verified 2023-04

CONDITIONS: Prosthetic Valve Endocarditis (PVE)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- endocarditis (Experimental)
  Interventions: Device: 18F-FDG PET/CT

INTERVENTIONS:
Device: 18F-FDG PET/CT

SUMMARY:
The diagnosis of prosthetic valve endocarditis (PVE) remains challenging. In PVE cases, initial echocardiography is normal or inconclusive in almost 30% of cases, leading to a decreased diagnostic accuracy for the modified Duke criteria.

Aims: The investigators sought to determine the value of 18F-fluorodeoxyglucose positron emission tomography/computed tomography (18F-FDG PET/CT) for diagnosing PVE.

Methods: In two referral French centers (Timone Hospial, Marseille and Georges Pompidou European Hospital, Paris), the investigators plan to include consecutive patients suspected of having PVE. All of the patients will be subjected to clinical, microbiological, and echocardiographic evaluation. Cardiac PET/CT will be performed at admission and the data analysis will be based on visual interpretation and quantitative measurement of FDG uptake (SUVmax). The final diagnosis will be defined according to the clinical and/or pathological modified Duke criteria determined during a 3-month follow-up (gold standard).

ELIGIBILITY:
Inclusion Criteria:

* unexplained persistent or recurrent fever >38°C;
* and/or unexplained increased serum C-reactive protein (CRP) level >10 mg/L; and/or positive blood cultures, independent of the echocardiographic analysis results;
* and/or positive serological testing for Coxiella burnetii, Bartonella spp., Mycoplasma pneumoniae, Legionella pneumophila, Aspergillus spp., or Tropheryma whipplei;
* and/or a mass or a new partial prosthetic valve dehiscence observed using echocardiography.

Exclusion Criteria:

* pregnancy,
* an inability to lie flat,
* a need for urgent cardiac surgery,
* hemodynamic instability,
* cardiac surgery <1 month ago,
* and a blood glucose level >1.8 g/L. Patients with a poor PET/CT image quality

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2014-02-05 (Actual); Primary Completion 2018-03-20 (Actual); Study Completion 2023-04-21 (Actual)

PRIMARY OUTCOMES:
the diagnosis of prosthetic valve infective endocarditis | 39months
  18F-fluorodeoxyglucose positron emission tomography

SECONDARY OUTCOMES:
the reproducibility of the technique, | 39 months
  the other diagnostic parameters of PET/CT (specificity and predictive values)
the comparison of the sensitivity of PET/CT with that of echocardiography, | 39 MONTHS
  the other diagnostic parameters of PET/CT (specificity and predictive values)
the rate of detection of embolic events, | 39 MONTHS
  the other diagnostic parameters of PET/CT (specificity and predictive values)
the prognostic value of the technique (death/valve surgery) | 39 MONTHS
  the other diagnostic parameters of PET/CT (specificity and predictive values)

CONTACTS AND LOCATIONS:
Overall Officials: LOIC MONDOLONI, Study Director — Assistance Publique Hopitaux De Marseille
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France